CLINICAL TRIAL: NCT04469452
Title: Validation of the Apollo EE Device, Indirect Calorimetry
Brief Title: Validation of a Portable Indirect Calorimeter
Status: Terminated | Type: Observational
Why Stopped: Halted by sponsor
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0317
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Human Energy Expenditure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adults (19-99yrs): Healthy adults already enrolled in separate studies using indirect calorimetry to measure RMR within our lab will be recruited for this study. Fifty participants (25 male, 25 female) will be heterogeneous in age, body composition, and physical activity based on the inclusion and exclusion of their respective studies. To test reliability, 25 of the 50 participants will repeat RMR measurements within 1 week of initial measurements.
  Interventions: Device: Apollo Device

INTERVENTIONS:
Device: Apollo Device — Comparisons will be made between the Apollo EE Device (Sable Systems International, Las Vegas, NV) and the TrueOne 2400 metabolic cart (Parvo Medics, Salt Lake City, UT)

SUMMARY:
This study plans to test the accuracy of a new device (the Apollo EE Device) that measures resting energy expenditure (REE) using only oxygen consumed (VO2). Findings from this study will help determine how this new device compares to the gold standard, indirect calorimetry, which measures REE using VO2 and carbon dioxide production (VCO2). Findings may help develop less expensive and more accessible means of measuring energy expenditure.

DETAILED DESCRIPTION:
The gold standard for measuring resting metabolic rate (RMR) is metabolic carts that measure oxygen consumption (VO2) and carbon dioxide production (VCO2). The energy equivalent of VO2 ranges from ~4.7-5.0 kcals/L, depending on the ratio of carbohydrate, fat, and protein oxidized. However, RMR can be measured based solely on VO2, because VCO2 has a relatively small effect on energy expenditure estimation. A device that measures RMR based on VO2 and eliminates the need for measuring VCO2 could provide a simple and less expensive alternative to metabolic carts and may have important clinical applications. The overarching goal of this proposal is to validate such a metabolic system by comparing its ability to accurately measure RMR against a metabolic cart.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 19-99 yrs of age

Exclusion Criteria:

* Pregnancy

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Only individuals who are enrolled in a separate study using indirect calorimetry to measure RMR within our lab will be eligible to participate in this study.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Accuracy of a new indirect calorimeter, the Apollo EE Device, when compared to the gold standard (TrueOne 2400 metabolic cart) | Baseline
  Measurement of RMR
Reliability of a new indirect calorimeter, the Apollo EE Device, when compared to the gold standard (TrueOne 2400 metabolic cart) | Repeated Measure obtained within 1 week of baseline measure
  Repeated measurement of RMR

CONTACTS AND LOCATIONS:
Overall Officials: Edward Melanson, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No